CLINICAL TRIAL: NCT04156672
Title: REal-world Study of the Clinical Profile and Treatment Outcomes of Advanced Therapies for Ulcerative Colitis in Portugal-READ UC
Brief Title: Real World Study Of The Clinical Profile And Treatment Outcomes Of Advanced Therapies For Ulcerative Colitis In Portugal
Acronym: READ-UC
Status: Withdrawn | Type: Observational
Why Stopped: Study was cancelled due to reclassification of study design. No subjects enrolled in the study.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A3921353; READ UC (Other: Alias Study Number)
Record Dates: First submitted 2019-10-24; First posted 2019-11-07 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional

SUMMARY:
This study aims to characterize the Portuguese population of patients with moderate-to-severe UC receiving advanced therapies, by describing clinical and sociodemographic characteristics, and remission outcomes . The clinical, biochemical, endoscopic, and histological outcomes will also be described, as well as frequency of selected EIM, comorbidities and the uptake of preventive care measures and hospitalizations .

ELIGIBILITY:
Inclusion Criteria:

* Aged at least 18 years old
* Diagnosed with Ulcerative Colitis, confirmed by a gastroenterologist
* Treated with anti-TNF or anti-integrin or JAK inhibitors drugs for at least 16 weeks
* Followed at one of the participating centers when initiating and during the current treatment
* Signed informed consent

Exclusion Criteria:

* Treated with anti-TNF or anti-integrin or JAK inhibitors drugs at induction phase
* Enrolled in randomized clinical trials or other experimental studies in the last 12 months prior to initiation of advanced therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients followed at Portuguese gastroenterology services, presenting moderate-to-severe Ulcerative Colitis and receiving advanced therapies (i.e., anti-TNF or anti-integrin or JAK inhibitors drugs) for at least 16 weeks.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-10-06 (Estimated); Primary Completion 2021-04-30 (Estimated); Study Completion 2021-04-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants achieving remission at study appointment, defined as both symptomatic and faecal biomarker remission | at baseline
  - percentage of participants with both a Mayo stool frequency subscore of 0 or 1 and Mayo rectal bleeding subscore of 0 , and a Faecal Calprotectin concentrations < to the cut-off concentration of 150-200 μg/g
Demographics and clinical characteristics of Ulcerative Colitis participants | till baseline
  * percentage of gender distribution, age distribution, smoking status distribution, height and weight distribution, BMI distribution
  * percentage of Ulcerative Colitis extend and severity (Montreal criteria) distribution, percentage of prior acute severe Ulcerative Colitis, percentage of clinical relapses

SECONDARY OUTCOMES:
Proportion of participants achieving remission at study appointment, defined as both symptomatic and faecal biomarker remission, by previous treatment line and by treatment duration | at baseline
Proportion of Ulcerative Colitis participants with symptomatic remission | at baseline
Duration of symptomatic remission | since initiation symptomatic remission till baseline
Proportion of participants with faecal biomarker <150-200 μg/g and >150-200 μg/g | at baseline
Proportion of participants with steroid use | at baseline
Total time without steroids since initiation of current advanced therapy | since initiation current advanced therapy till baseline
Proportion of participants in steroid-free remission | at baseline
Time spent in hospital, including all Inflammatory Bowel Disease-related admissions requiring an overnight stay | since initiation current advanced therapy till baseline
Frequency and incidence of hospitalizations and emergency visits | since initiation current adavnced therapy till baseline
Frequency of registered preventive care measures | in the 12 months prior initiation current advanced therapy till baseline
Proportion of Ulcerative Colitis participants with history or current evidence of Extra Intestinal Manifestations | till baseline
Proportion of Ulcerative Colitis participants with history or current evidence of comorbidities | till baseline

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.